CLINICAL TRIAL: NCT02475460
Title: Thoratec Corporation HeartMate 3™ Less Invasive Surgery (LIS) Study
Brief Title: HeartMate 3™ LIS Study
Acronym: HM 3 LIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Thoratec Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HeartMate 3 LIS
Record Dates: First submitted 2015-06-11; First posted 2015-06-18 (Estimated); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Heart Failure; Cardiovascular Disease
Keywords: HeartMate 3; LVAS; LVAD; Heart-assist Devices; Advanced; Ventricular Dysfunction; refractory left ventricular; Thoratec Corporation
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases; Ventricular Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HM 3 LIS (Experimental): All patients implanted with the HM 3 LVAD via less invasive surgical technique
  Interventions: Procedure: Less Invasive Surgery (LIS); Device: HeartMate 3™

INTERVENTIONS:
Procedure: Less Invasive Surgery (LIS) — Less invasive HM 3 LVAD surgical implant procedure
Device: HeartMate 3™ — HM 3 LIS

SUMMARY:
The purpose of this study is to evaluate a less invasive implantation technique of the HeartMate 3 Left Ventricular Assist System (HM 3 LVAS) in 10 patients.

DETAILED DESCRIPTION:
This study will evaluate the less invasive implantation technique of the HM 3 LVAS.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or legal representative has signed Informed Consent Form (ICF)
2. Age ≥ 18 years
3. BSA ≥ 1.2 m2
4. NYHA IIIB or IV, or ACC/AHA Stage D
5. LVEF ≤ 25%
6. CI ≤ 2.2 L/min/m2, while not on inotropes (if Patient is treated with inotropes at baseline, this does not apply)
7. Patients must also meet one of the following:

   * On optimal medical management (OMM), based on current heart failure practice guidelines for at least 45 out of the last 60 days and are failing to respond, OR
   * In NYHA class IIIB or IV heart failure for at least 14 days AND dependent on intraaortic balloon pump (IABP) for at least 7 days, OR
   * Inotrope dependent/unable to wean from inotropes OR
   * Listed for transplant
8. Females of child bearing age must agree to use adequate contraception-

Exclusion Criteria:

1. Etiology of heart failure (HF) due to or associated with uncorrected thyroid disease, obstructive cardiomyopathy, pericardial disease, amyloidosis or restrictive cardiomyopathy
2. Technical obstacles which pose an inordinately high surgical risk, in the judgment of the Investigator
3. Existence of ongoing mechanical circulatory support (MCS) other than IABP
4. Positive pregnancy test if of childbearing potential
5. Lactating mothers
6. Presence of mechanical aortic cardiac valve
7. History of any organ transplant
8. Platelet count < 100,000 x 103/L (< 100,000/ml)
9. Psychiatric disease/disorder, irreversible cognitive dysfunction or psychosocial issues that are likely to impair compliance with the study protocol and LVAS management
10. History of confirmed, untreated AAA > 5 cm in diameter
11. Presence of an active, uncontrolled infection
12. Intolerance to anticoagulant or antiplatelet therapies or any other peri/post-operative therapy that the Investigator will require based upon the patients' health status
13. Presence of any one of the following risk factors for indications of severe end organ dysfunction or failure:

    * An INR ≥ 2.5 not due to anticoagulation therapy
    * Total bilirubin > 43 umol/L (2.5 mg/dl), shock liver, or biopsy proven liver cirrhosis
    * History of severe chronic obstructive pulmonary disease (COPD) defined by FEV1/FVC < 0.7, or FEV1 <50% predicted
    * Fixed pulmonary hypertension with a most recent PVR ≥ 8 Wood units that is unresponsive to pharmacologic intervention
    * History of stroke within 90 days prior to enrollment, or a history of cerebrovascular disease with significant (> 80%) carotid artery stenosis
    * Serum Creatinine ≥ 221umol/L (2.5 mg/dl) or the need for chronic renal replacement therapy
    * Significant peripheral vascular disease (PVD) accompanied by rest pain or extremity ulceration
14. Aortic valve regurgitation > grade 1
15. Pre albumin < 150 mg/L, or Albumin < 30g/L (3 g/dL)
16. Planned Bi-VAD support prior to enrollment
17. Patient has known hypo or hyper coagulable states such as disseminated intravascular coagulation and heparin induced thrombocytopenia
18. Planned concomitant intra-cardiac cardiac surgery
19. Thrombus formation in the atrium or left ventricle identified by echocardiogram
20. Previous sternotomy or left-sided thoracotomy
21. Participation in any other clinical investigation that is likely to confound study results or affect the study
22. Any condition other than HF that could limit survival to less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of survival participants | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Sami Somo, Study Director — Abbott
Locations (3):
- Institute for Clinical and Experimental Medicine (IKEM), Prague, Czechia
- Germany (2):
  - Deutsches Herzzentrum Berlin, Berlin
  - Medizinische Hochschule Hannover, Hanover